CLINICAL TRIAL: NCT07144384
Title: A Pilot Study Testing Intralesional Injection of Ex-Vivo Expanded Allogenic University Donor (UD) NK and TGFBi NK Cells in Patients With Cutaneous Keratinocyte Carcinomas
Brief Title: Intratumoral Injection of Standard Universal Donor Expanded Natural Killer Cells and TGF-beta Imprinted Natural Killer Cells for the Treatment of Skin Squamous Cell Carcinoma and Basal Cell Carcinoma
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Brittany Dulmage (Other)
Responsible Party: Sponsor-Investigator, Brittany Dulmage, Principal Investigator, Ohio State University Comprehensive Cancer Center
Organization: Ohio State University Comprehensive Cancer Center (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OSU-24311; NCI-2025-05655 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2025-08-12; First posted 2025-08-27 (Actual); Last update posted 2025-10-24 (Actual); Status verified 2025-10

CONDITIONS: Skin Basal Cell Carcinoma; Skin Nodular Basal Cell Carcinoma; Skin Squamous Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Basal Cell | interventions — Biopsy; Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cohort I (UD expanded NK cells) (Experimental): Patients undergo SOC biopsy on day 0 and within 4 weeks (days 10-28) receive UD expanded NK cells intratumorally. Patients undergo SOC excision 4-8 weeks (days 28-56) after biopsy.
  Interventions: Procedure: Biopsy Procedure; Biological: Natural Killer Cell Therapy; Procedure: Surgical Procedure
- Cohort II (UD expanded TGFbetai NK cells) (Experimental): Patients undergo SOC biopsy on day 0 and within 4 weeks (days 10-28) receive UD expanded TGF-beta-i NK cells intratumorally. Patients undergo SOC excision 4-8 weeks (days 28-56) after biopsy.
  Interventions: Procedure: Biopsy Procedure; Procedure: Surgical Procedure; Biological: Universal Donor Expanded TGF-beta-imprinted NK Cells

INTERVENTIONS:
Procedure: Biopsy Procedure — Undergo SOC biopsy
  Other Names: Biopsy; BIOPSY_TYPE; Bx
Biological: Natural Killer Cell Therapy — Given UD expanded NK cells intratumorally
  Arms: Cohort I (UD expanded NK cells)
Procedure: Surgical Procedure — Undergo SOC excision
  Other Names: Operation; Surgery; Surgery Type; Surgery, NOS; Surgical; Surgical Intervention; Surgical Interventions; Surgical Procedures; Type of Surgery
Biological: Universal Donor Expanded TGF-beta-imprinted NK Cells — Given intratumorally
  Other Names: Allogeneic TGFBi Expanded NK Cells; UD TGF-betai NK Cells; Universal Donor TGF-beta Imprinted Expanded NK Cells
  Arms: Cohort II (UD expanded TGFbetai NK cells)

SUMMARY:
This early phase I trial compares the safety, side effects and the biological or cellular activity of two types of universal donor (UD) natural killer (NK) cells (standard NK cells and transforming growth factor [TGF] beta imprinted [TGF-beta-i] NK cells), given directly into the tumor (intratumoral) in treating patients with skin (cutaneous) squamous cell carcinoma (SCC) or basal cell carcinoma (BCC). NK cells are a type of white blood cell that can recognize missing or incorrect proteins on tumor cells and then kill these tumor cells. It was recently discovered that infection with human cytomegalovirus (CMV), a common virus, leads to the development of a unique NK cell population. These "adaptive" NK cells have a more potent anti-tumor killing action. The TGF-beta-i NK cells used in this study are created using donors whose blood tests positive for CMV exposure. This may make them more effective at killing tumor cells. Giving UD TGF-beta-i NK cells may be safe, tolerable and/or more effective than standard UD expanded NK cells in treating patients with SCC or BCC.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine the persistence of NK cell infiltration within biopsy-proven keratinocyte carcinomas following intra-tumoral injection of universal donor NK cells versus (vs) TGFbeta-resistant NK cells in a cohort of patients prior to their standard of care excision.

SECONDARY OBJECTIVES:

I. To assess the tolerability of NK cell cutaneous intra-tumoral injection measured by adverse events, described using Common Terminology for Cancer Related Adverse Events (CTCAE version [v] 5).

II. To test the feasibility of a larger study using intra-tumorally injected NK cells.

EXPLORATORY/CORRELATIVE OBJECTIVES:

I. To assess clinical outcomes including size, area change, and visual appearance in clinical detection of keratinocyte carcinomas between injection and excision.

II. To compare NK and other immune cell presence within the tumor/tumor microenvironment (TME) in cutaneous basal cell carcinomas (BCCs) vs squamous cell carcinomas (SCCs) injected with NK vs TGFbetai cells prior to excision.

OUTLINE: Patients are randomized to 1 of 2 cohorts.

COHORT I: Patients undergo standard of care (SOC) biopsy on day 0 and within 4 weeks (days 10-28) receive UD expanded NK cells intratumorally. Patients undergo SOC excision 4-8 weeks (days 28-56) after biopsy.

COHORT II: Patients undergo SOC biopsy on day 0 and within 4 weeks (days 10-28) receive UD expanded TGF-beta-i NK cells intratumorally. Patients undergo SOC excision 4-8 weeks (days 28-56) after biopsy.

ELIGIBILITY:
Inclusion Criteria:

* Ohio State University patients > 18 years old
* Diagnosis of ≥ 1cm keratinocyte carcinoma, accessible by intra-tumoral injection
* Confirmation of cutaneous SCC (cSCC) (10 patients total) or BCC (10 patients total) via diagnostic biopsy

  * BCC: Nodular or aggressive subtype
  * SCC: Well-differentiated or aggressive subtype with T1 or T2 staging by American Joint Committee on Cancer (AJCC) criteria
* Patient meets criteria for standard of care surgical treatment with either wide local excision or Moh's surgery
* Presence of residual clinical cancer ≥ 1cm at the time of baseline
* Willingness to follow up for residual cancer extirpation between 2-8 weeks after the injection

Exclusion Criteria:

* Planned or concurrent radiation or systemic treatment for solid tumor or hematologic malignancy including chemotherapies or immunotherapies received within 6 weeks of trial enrollment. These include but are not limited to methotrexate, 5-fluorouracil, vismodegib, cepilimumab, pembrolizumab, nivolumab, ipilimumab for any skin malignancy
* < 18 years old
* A negative deep and peripheral margin status from the diagnostic biopsy
* Diagnostic biopsy with the following histopathologic characteristics:

  * BCC: Superficial subtype
  * SCC: SCC in situ (SCCIS)/Bowen disease, basosquamous, keratoacanthoma (KA)-type SCC, or tumor with > T2 staging by AJCC criteria
* Any skin disease or active infection in the same area that may confound assessments
* Inability to follow-up for definitive treatment (surgical excision)
* Any other comorbidity or complication that in the opinion of the investigator could make the patient unsafe to participate in the study, such as:

  * Active infection
  * Pregnant women, women who are likely to become pregnant or are breastfeeding
  * Patients who received any other investigational drugs within the 30 days prior to screening visit

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-10-16 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in intratumoral natural killer (NK) cell content | Up to 2 weeks after locoregional injection of NK cells
  Immunohistochemical and in vitro studies of tissue from the original biopsy and post-NK cell treated tumor specimens will be performed to assess NK cell infiltration of the tumor. Difference in NK cell density by CD56 staining in pre- versus post-intervention skin tumor tissue will be compared between tumors receiving NK versus transforming growth factor betai cell injections.

SECONDARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by Common Terminology Criteria for Adverse Events version 5.0 criteria | Up to 8 weeks after biopsy
  Will be assessed by Common Terminology Criteria for Adverse Events version 5.0 criteria. Will be summarized as the percentage of patients experiencing each type and grade of event according to dose level. Frequency and severity of AEs and tolerability of the regimen will be collected and summarized by descriptive statistics. The maximum grade for each type of toxicity will be recorded for each patient, and frequency tables will be reviewed to determine toxicity patterns.

CONTACTS AND LOCATIONS:
Overall Officials: Brittany L Dulmage, MD, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (1):
- Ohio State University Comprehensive Cancer Center, Columbus, Ohio, United States

REFERENCES:
- See also: The Jamesline — http://cancer.osu.edu